CLINICAL TRIAL: NCT05892562
Title: A Causal Relationship Study Between Anxiety, Depression, and Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shate Xiang (Other Government)
Collaborators: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor-Investigator, Shate Xiang, Principal Investigator, Zhejiang Chinese Medical University
Organization: Zhejiang Chinese Medical University (Other Government)
Other Study IDs: Shate Xiang
Record Dates: First submitted 2023-04-19; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Rheumatoid Arthritis; Anxiety; Depression
MeSH Terms: conditions — Arthritis, Rheumatoid; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RA combined with depression or anxiety
  Interventions: Other: No intervention
- RA without comorbid depression or anxiety
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — As this study is purely observational, no intervention is involved.

SUMMARY:
Rheumatoid arthritis (RA) is a systemic chronic inflammatory disease, and depression and anxiety are among the most common comorbidities in RA patients, with a high prevalence rate. Epidemiological studies have found that joint deformities, severe pain, positive serum RF titers, as well as comorbidities such as hypertension, insomnia, pain, and fatigue are significantly associated with depression and anxiety in RA patients.

Currently, clinical studies have found that the relief of depression or anxiety is one of the expected treatment goals for RA patients. Due to the unclear pathogenic factors of depression or anxiety in RA patients, there is a lack of effective clinical treatment options. Therefore, this study will use a "causal inference model" to identify possible "mediating variables" that may lead to the comorbidity of RA and emotional disorders through clinical investigation, aiming to improve the precision of treatment for physicians.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with RA.

Exclusion Criteria:

* Patients diagnosed as non-RA.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Our study population consists of patients diagnosed with RA in clinical settings, who were assessed for their mental status using PHQ-9 and GAD-7, and classified as either RA patients with comorbid depression or RA patients without comorbid depression.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Enrollment: January 2022 to May 2023
  The PHQ-9, one of the internationally recognized depression screening tools, consists of 9 items that correspond to common symptoms of depression, including depressed mood, loss of interest, sleep problems, fatigue, changes in appetite, self-evaluation issues, concentration difficulties, psychomotor problems, and suicidal thoughts. Each item has four response options representing the frequency or severity of symptoms, including "0" (not at all), "1" (several days), "2" (more than half the days), and "3" (nearly every day). By summing the scores of these 9 items, a total score is obtained to measure the severity of depression. The total score ranges from 0 to 27, with higher scores indicating greater severity of depressive symptoms.
Generalized Anxiety Disorder-7 (GAD-7) | Enrollment: January 2022 to May 2023
  The GAD-7 scale is a commonly used self-assessment tool to evaluate the severity of generalized anxiety disorder. It consists of 7 items that correspond to common symptoms of generalized anxiety disorder, including excessive worry, nervousness, anxiety, irritability, difficulty concentrating, fatigue, and muscle tension. Similar to the PHQ-9, each item has four response options representing the frequency or severity of symptoms. The response options include "0" (not at all), "1" (several days), "2" (more than half the days), and "3" (nearly every day). By summing the scores of these 7 items, a total score is obtained to measure the severity of generalized anxiety disorder. The total score ranges from 0 to 21, with higher scores indicating greater severity of anxiety symptoms.

SECONDARY OUTCOMES:
Body Mass Index | Enrollment: January 2022 to May 2023
  The Body Mass Index (BMI) is a commonly used measure of body weight in relation to height. It is calculated by dividing a person's weight in kilograms by the square of their height in meters. The formula for calculating BMI is:
  BMI = weight (kg) / height (m)^2
  Based on the calculated value, BMI categorizes individuals into different weight ranges. The commonly used classification criteria are as follows:
  BMI < 18.5: Underweight 18.5 ≤ BMI < 24.9: Normal weight 25 ≤ BMI < 29.9: Overweight BMI ≥ 30: Obesity
Marital status | Enrollment: January 2022 to May 2023
  We categorized the marital status of the study population into three major groups: married, unmarried, and divorced.
Educational level | Enrollment: January 2022 to May 2023
  We categorized the educational level of the study population into three categories: primary school or below, junior high school or high school, and college or above.
Financial status | Enrollment: January 2022 to May 2023
  We classified the patients' satisfaction with their current economic situation into three categories: comfortable, manageable, and challenging.
Smoking history | Enrollment: January 2022 to May 2023
  Smoking history: Never smoked, Former smoker, Current smoker.
Disease Activity Score 28 | Enrollment: January 2022 to May 2023
  DAS28 (Disease Activity Score 28) is a scale used to assess the activity level of rheumatoid arthritis (RA). It is calculated based on the assessment of joint swelling, joint tenderness, systemic inflammatory markers (erythrocyte sedimentation rate), and the patient's self-assessment of pain using a visual analog scale (VAS). The specific formula for calculating DAS28 (Disease Activity Score 28) is as follows:
  DAS28 = 0.56 * √(TJC28) + 0.28 * √(SJC28) + 0.36 * ln(CRP) + 0.014 * GH + 0.96 The DAS28 calculation includes the examination of 28 joints, including the fingers and wrists, elbows, shoulders, knees, and ankles. The DAS28 score ranges from 0 to 10, with higher scores indicating higher disease activity. Common classification criteria include low disease activity (DAS28 < 3.2), moderate disease activity (3.2 ≤ DAS28 < 5.1), and high disease activity (DAS28 ≥ 5.1).
Labor intensity based on the 2000 Chinese Nutrition Society's classification standard | Enrollment: January 2022 to May 2023
  Light physical activity: Refers to activities such as prolonged standing or walking, office work, light household chores, etc.
  Moderate physical activity: Refers to activities that involve more walking, standing work, moderate household chores, farming, and light physical work.
  Heavy physical activity: Refers to activities such as prolonged walking or running, heavy physical work, sports athletes, and other high-intensity activities.
Health Assessment Questionnaire Disability Index (HAQ-DI) | Enrollment: January 2022 to May 2023
  The Health Assessment Questionnaire Disability Index (HAQ-DI) is a commonly used scale for assessing the level of functional disability in patients' daily activities. It covers various activities such as getting up, dressing, bathing, eating, walking, and climbing stairs. Patients are required to rate each item based on their actual abilities to reflect their level of functional impairment. The scoring typically ranges from 0 to 3, with 0 indicating no functional disability and 3 indicating severe functional impairment.The minimum value is 0, and the maximum value is 60.
  By calculating the total score of HAQ-DI, the quantified assessment of patients' daily life functioning can be obtained. This index can be used to evaluate treatment effectiveness, disease progression, and quality of life changes in patients.
  Note that HAQ-DI is not only used for assessing patients with rheumatoid arthritis but can also be applied to functional assessment in other chronic diseases.
The Fatigue Self-Assessment Scale. | Enrollment: January 2022 to May 2023
  The Fatigue Self-Assessment Scale (FSAS) is developed based on a review of research on fatigue assessment both domestically and internationally, taking into account Chinese language habits and cultural characteristics. The scale consists of 23 items and is used to assess the types and severity of fatigue in sub-healthy individuals and various patient populations with fatigue-related symptoms. It includes three factors: physical fatigue, mental fatigue, and consequences of fatigue. It also evaluates three characteristics of fatigue: response to sleep/rest, situational factors, and temporal patterns. The scale can be used to assess the effectiveness of interventions targeting fatigue. The minimum score is 0, and the maximum score is 88, with higher scores indicating greater levels of fatigue.
The Pittsburgh Sleep Quality Index (PSQI) | Enrollment: January 2022 to May 2023
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire used to assess an individual's sleep quality and disturbances over a one-month time period. It consists of 19 items that cover several aspects of sleep, including sleep duration, sleep latency, sleep disturbances, use of sleep medications, and daytime dysfunction. The questionnaire is scored on a 0 to 3 scale for each item. The total score ranges from 0 to 21, with a higher score indicating worse sleep quality. The PSQI is commonly used in research and clinical settings to evaluate sleep problems and monitor treatment outcomes.
Complications | Enrollment: January 2022 to May 2023
  For example, hypertension, diabetes, Sjogren's syndrome, etc. We do not document diseases that have been treated with surgical procedures, such as uterine fibroids that have been removed.
Medication use | Enrollment: January 2022 to May 2023
  Mainly record the medication used by patients to treat rheumatoid arthritis in the past half month. For example, methotrexate, leflunomide, hydroxychloroquine, etc
Alcohol history | Enrollment: January 2022 to May 2023
  Alcohol history: Never drank, Former drinker, Current drinker.
Surgical history | Enrollment: January 2022 to May 2023
  Surgical history: No history of surgery, History of surgery.
Erythrocyte sedimentation rate (mm/h) | Enrollment: January 2022 to May 2023
  Erythrocyte sedimentation rate (ESR) is a blood test that measures the rate at which red blood cells settle in a vertical tube over a specific period of time. It is a non-specific marker of inflammation and is commonly used as a screening test to assess the presence and severity of inflammatory conditions in the body.
White blood cell count (cells/μL) | Enrollment: January 2022 to May 2023
  White blood cell count, also known as leukocyte count, is a blood test that measures the number of white blood cells (leukocytes) present in a specified volume of blood. White blood cells are an essential part of the immune system.
Anti-nuclear antibodies | Enrollment: January 2022 to May 2023
  When the test result is negative or 1:20, we consider it negative. When the result is 1:40, we consider it weakly positive. When the result is 1:60 or higher, we consider it positive.
Anti-cyclic citrullinated peptide antibody (U/mL) | Enrollment: January 2022 to May 2023
  Anti-cyclic citrullinated peptide antibody (anti-CCP antibody) is a type of autoantibody that targets the synthetic cyclic citrullinated peptide (CCP) antigen. It has high sensitivity and specificity for rheumatoid arthritis (RA), making it a highly specific marker for early diagnosis of RA. Furthermore, patients who test positive for this antibody are more likely to develop severe joint damage compared to those who test negative for the antibody.
Hypersensitive C-reactive protein (mg/L) | Enrollment: January 2022 to May 2023
  Hypersensitivity C-reactive protein (hsCRP) is a highly sensitive blood biomarker for measuring C-reactive protein levels. It is measured in milligrams per liter (mg/L). The level of hsCRP in the blood reflects the level of inflammation in the body.
Rheumatoid factor (IU/ml) | Enrollment: January 2022 to May 2023
  Rheumatoid factor (RF) is an autoantibody that targets the Fc portion of immunoglobulin G (IgG) antibodies. It is measured in international units per milliliter (IU/ml). Elevated levels of RF in the blood are commonly associated with rheumatoid arthritis (RA) and other autoimmune conditions. The presence of RF in the blood indicates an immune system response and can contribute to the diagnosis and management of RA.

OTHER OUTCOMES:
weight | Enrollment: January 2022 to May 2023
  weight in kilograms
height | Enrollment: January 2022 to May 2023
  height in meters
Visual Analogue Scale | Enrollment: January 2022 to May 2023
  VAS (Visual Analog Scale) is a pain assessment scale that uses a ruler divided into 10 equal parts. A score of 0 represents no pain, while a score of 10 represents the highest level of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, None Selected, China

IPD SHARING:
Plan to Share IPD: No